CLINICAL TRIAL: NCT04265573
Title: Feasibility, Acceptability and Costs of a Strategy Deploying Multiple First-lines Artemisinin-based Combination Therapies for Uncomplicated Malaria: a Pilot Programme in the Health District of Kaya, Burkina Faso
Brief Title: Feasibility, Acceptability and Costs of a Multiple First-lines Artemisinin-based Combination Therapies
Status: Completed | Type: Observational
Sponsor: Groupe de Recherche Action en Sante (Other)
Collaborators: Medicines for Malaria Venture (Other); National Malaria Control Programme (NMCP), Burkina Faso (Unknown); Institut de Recherche en Sciences de la Sante, Burkina Faso (Other Government)
Responsible Party: Sponsor
Other Study IDs: MFTs-ACTs-BF (PO17/01110)
Record Dates: First submitted 2020-01-21; First posted 2020-02-11 (Actual); Last update posted 2022-03-25 (Actual); Status verified 2020-02

CONDITIONS: Malaria
Keywords: Uncomplicated malaria; Multiple First-lines Therapies; Artemisinin-based Combination Therapy; Acceptability; Feasability; Costs
MeSH Terms: conditions — Malaria

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Children under-five: Uncomplicated malaria case in this group will be managed using Pyronaridine-Artesunate at health facility level. This drug is registered in Burkina Faso for routine medical care for uncomplicated malaria case.
- Individuals five years of age and above: Uncomplicated malaria case in this group will be managed using Dihydoartemisinin-Piperaquine health facility level. This drug is registered in Burkina Faso for routine medical care for uncomplicated malaria case.
- Pregnant women: Uncomplicated malaria case in this group will be managed using Artemether-Lumefantrin health facility level. This drug is registered in Burkina Faso for routine medical care for uncomplicated malaria case.

SUMMARY:
A simultaneous deployment of multiple first line therapies (MFT) for uncomplicated malaria using artemisisin based combination therapies as showed by theoretical models, may extend the useful therapeutic life of the current Artemisinin-based combination thérapies (ACTs) by reducing drug pressure and slowing the spread of resistance without putting life at risk. We therefore hypothesized that a simultaneous deployment of three ACTs targeting three segments of the population is feasible, acceptable and can achieve high coverage rate if potential barriers are well identified, well addressed and the key implementers are well-trained and adequately supported. To test this hypothesis, a quasi-experimental study will be conducted.

DETAILED DESCRIPTION:
The study will be conducted through four overlapping phases: formative research phase, the MFTs deployment phase, the evaluation phase and the post-evaluation phase.

1. Formative research phase

   1.1 Objective

   Generate baseline information and to develop intervention tools for the pilot implementation of MFTs for uncomplicated malaria in the study area.

   1.2 Design

   Cross-sectional surveys using desk reviews, qualitative and quantitative research methods:
   * Individual in-depth Interviews
   * Focus group discussions
   * Household surveys for the assessment of malaria-related morbidity and mortality at community level as well as the healthcare system utilisation
   * Health facility-based surveys for malaria morbidity and mortality, antimalarial drugs and malaria rapid diagnostic tests availability.

   1.3 Duration

   Six months from obtaining the approval of the ethics committee for health research.
2. MFTs deployment phase

   2.1 Objective

   Implement the MFTs for uncomplicated malaria in the health district of Kaya that is feasible, acceptable and achieve high coverage rate.

   2.2 Drugs deployment

   Study ACTs and respective target populations:
   * Artesunate-Pyronaridine for children less than five years of age
   * Artemether-Lumefantrine for pregnant women
   * Dihydroartemisinin-Piperaquine for individuals five years of age and above

   NB: Community case management of malaria using Artemether-Lumefantrine as per National Malaria Control Program recommendation.

   2.3 Duration

   Twelve months including low and high malaria transmission seasons in the study area.
3. Monitoring and evaluation phase

   3.1 Objectives

   Assess the feasibility, the acceptability, the cost and the effects of the pilot MFTs pilot programme for uncomplicated malaria in the health district of Kaya.

   3.2 Design

   Cross-sectional surveys using desk review, qualitative and quantitative research methods:
   * Individual in-depth Interviews
   * Focus group discussions
   * Household surveys for the assessment of malaria-related morbidity and mortality at community level as well as the healthcare system utilisation
   * Health facility-based surveys for malaria-related morbidity and mortality, the availability and use of antimalarial drugs and malaria rapid diagnostic tests.
   * Costs assessments.

   3.3 Duration

   Four months.
4. Post-evaluation phase

4.1 Objectives

Communicating and disseminating the findings of the pilot implementation of multiple first-lines artemisinin-based combination therapies for uncomplicated malaria in the health district of Kaya, Burkina Faso;

4.2 Methodology

* Feedback meetings for reporting to local communities
* National workshop aiming at reporting the programme findings
* Final report to be submitted to the donor
* Oral presentations of findings at congresses, conferences, seminars and publication of findings in peer-reviewed scientific journals

ELIGIBILITY:
Inclusion Criteria:

Household survey

* Caregivers, adults, pregnant women
* Signed consent form

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The target populations for the deployment of the MFTs for uncomplicated malaria are: children less than five years of age, pregnant women, individuals five years of age and above.
Sampling Method: Non-Probability Sample
Enrollment: 150000 (Actual)
Dates: Start 2018-11-10 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2021-02-25 (Actual)

PRIMARY OUTCOMES:
Number of favourable and unfavourable opinions from various profiles of informants about the MFT pilot program. | From the formative phase to the end of drugs deployment: 18 months duration.
  Data will be collected through qualitative surveys (FGDs; IDIs) and quantitative households surveys (KAP questionnaire) from various profiles of informants.

SECONDARY OUTCOMES:
Proportion of community resources people with favourable opinions to the MFTs pilot program. | From the formative phase to the end of drugs deployment: 18 months duration.
  Data will be collected at community level through qualitative surveys (FGDs; IDIs) from various profiles of informants.
Proportion of community resources people with unfavourable opinions to the MFTs pilot program. | From the formative phase to the end of drugs deployment: 18 months duration.
  Data will be collected at community level through qualitative surveys (FGDs; IDIs) from various profiles of informants.
Average number of monitoring visits performed per annum | Through the MFTs deployment phase: 12 months of duration.
  Data will be obtained though the health facility- based surveys.
Average number of monitoring visits on which drugs stores have stock out of any dose of study ACTs per annum. | Through the MFTs deployment phase: 12 months of duration.
  Data will be obtained though the health facility- based surveys.
Average number of monitoring visits on which health facilities have stock out of mRDTs per annum. | Through the MFTs deployment phase: 12 months of duration.
  Data will be obtained though the health facility- based surveys.
Proportion of febrile episode seen at health facility level. | Through the MFTs deployment phase: 12 months of duration
  Data will be obtained through health facility- based surveys using registers of Health Facilities (HF).
Proportion of febrile episode seen at health facility level (HFL) within 24 hours | Through the MFTs deployment phase: 12 months of duration
  Data will be obtained through health facility- based surveys using registers of HF.
Proportion of febrile episode seen at HFL within 24 hours and tested for parasitemia. | Through the MFTs deployment phase: 12 months of duration.
  Malaria diagnosis will done using malaria rapid diagnosis test (mRDT). Data will be obtained through health facility- based surveys using registers of HF.
Proportion of febrile episode seen at HFL within 24 hours with positive diagnostic test who were given ACT according to the MFTs strategy | Through the MFTs deployment phase: 12 months of duration.
  Malaria diagnosis will done using malaria rapid diagnosis test (mRDT). Data will be obtained through health facility- based surveys using registers of HF.
Proportion of febrile episode seen at HFL within 24 hours with negative diagnostic test who did not received any antimalarial. | Through the MFTs deployment phase: 12 months of duration.
  Malaria diagnosis will done using malaria rapid diagnosis test (mRDT). Data will be obtained through health facility- based surveys using registers of HF.
Proportion of febrile episode seen at HFL within 24 hours with negative diagnostic test who received an ACT. | Through the MFTs deployment phase: 12 months of duration.
  Malaria diagnosis will done using malaria rapid diagnosis test (mRDT). Data will be obtained through health facility- based surveys using registers of HF.
Proportion of febrile episodes treated with ACTs adhering to ACT treatment schedule (timing and doses) by HWs according to MFTs strategy | During MFTs deployment phase at peak malaria season: 6 months of duration.
  Household surveys (data will be collected in the community level through the KAP questionnaire).
Cost per additional febrile episode receiving prompt treatment or confirmed negative diagnosis | Through the MFTs deployment phase: 12 months of duration.
  Data will be obtained using the cost data collection forms through health facility- based surveys.
Cost per additional inappropriate antimalarial treatment avoided. | Through the MFTs deployment phase: 12 months of duration.
  Data will be obtained using the cost data collection forms through health facility- based surveys.
The cost per additional febrile episode appropriate managed for malaria with confirmed diagnosis | Through the MFTs deployment phase: 12 months of duration
  Data will be obtained using the cost data collection forms through health facility- based surveys.
The total cost per capita of intervention (provider perspective) | Through the MFTs deployment phase: 12 months of duration
  Data will be obtained using the cost data collection forms through health facility- based surveys.
The total cost per capita of intervention (societal perspective) | Through the MFTs deployment phase: 12 months of duration
  Data will be obtained using the cost data collection forms through household surveys (costing questionnaire administered at community level).
Cost to the HWs to participate to the MFTs strategy. | Through the MFTs deployment phase: 12 months of duration.
  Data will be obtained using the cost data collection forms through at health facilities level.
Proportion of episode of uncomplicated fever seen by HWs tested for malaria parasitemia. | From the formative phase to the end of drugs deployment: 18 months duration.
  Data will be obtained through the health facility- based surveys (data collected at health facilities level using the registers of HF).
Proportion of uncomplicated fever episodes/malaria seen by HW, tested positive and treated with correct dose of ACT according to MFTs pilot program | From the formative phase to the end of drugs deployment: 18 months duration.
  Data will be obtained through the health facility- based surveys (data collected at health facilities level using the registers of HF).
Proportion of febrile episodes treated with ACTs according to MFTs pilot programme by HWs provided with appropriate dosing advice | From the formative phase to the end of drugs deployment: 18 months duration.
  Data will be obtained through the health facility- based surveys (data collected at health facilities level using the registers of HF).
Proportion of uncomplicated febrile episodes/malaria seen by HWs provided with advice on danger signs. | From the formative phase to the end of drugs deployment: 18 months duration.
  Data will be obtained through the health facility- based surveys (data collected at health facilities level using the registers of HF).
Incidence of uncomplicated febrile episode/malaria within 4 weeks preceding the surveys | From the formative phase to the end of drugs deployment: 18 months duration.
  Household surveys before and during the MFTs deployment using KAP questionnaire administered at the community level.
Proportion of uncomplicated febrile episode/malaria seen at health facility level before and during the MFTs deployment in the study area. | Through the MFTs deployment phase: 12 months of duration.
  Data will be obtained through the health facility- based surveys (data collected at the health facility level using the registers of HF).
Mortality rate related to febrile episode/malaria before and during the pilot MFTs deployment. | From the formative phase to the end of drugs deployment: 18 months duration.
  Data will be collected through the Health and demographic surveillance system mortality data and health facility- based surveys (data collected at the health facility level using the registers of HF).
Proportion of individuals with fever in the last four weeks for whom advice or treatment was sought | From the formative phase to the end of drugs deployment: 18 months duration.
  Household surveys using KAP questionnaire administered at the community level
Proportion of individuals with fever in the last four week who sought treatment at HFL within 24 hours | From the formative phase to the end of drugs deployment: 18 months duration.
  Household surveys using KAP questionnaire administered at the community level.
Source of advice or care for those suffering from fever in the last four weeks | From the formative phase to the end of drugs deployment: 18 months duration.
  Household survey using KAP questionnaire administered at the community level.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamadou Siribié, MD, PhD, Principal Investigator — Groupe de Recherche Action en Sante; André-Marie Tchouatieu, MD, Principal Investigator — Medicine for Malaria Venture (MMV)
Locations (1):
- Groupe de Recherche Action en Santé, Ouagadougou, Burkina Faso

REFERENCES:
- [Result] Boni MF, White NJ, Baird JK. The Community As the Patient in Malaria-Endemic Areas: Preempting Drug Resistance with Multiple First-Line Therapies. PLoS Med. 2016 Mar 29;13(3):e1001984. doi: 10.1371/journal.pmed.1001984. eCollection 2016 Mar. PMID 27022739
- [Result] Boni MF, Smith DL, Laxminarayan R. Benefits of using multiple first-line therapies against malaria. Proc Natl Acad Sci U S A. 2008 Sep 16;105(37):14216-21. doi: 10.1073/pnas.0804628105. Epub 2008 Sep 9. PMID 18780786
- [Derived] Kabore JMT, Siribie M, Hien D, Soulama I, Barry N, Nombre Y, Dianda F, Baguiya A, Tiono AB, Burri C, Tchouatieu AM, Sirima SB. Attitudes, practices, and determinants of community care-seeking behaviours for fever/malaria episodes in the context of the implementation of multiple first-line therapies for uncomplicated malaria in the health district of Kaya, Burkina Faso. Malar J. 2022 May 30;21(1):155. doi: 10.1186/s12936-022-04180-z. PMID 35637506
- [Derived] Siribie M, Tchouatieu AM, Soulama I, Kabore JMT, Nombre Y, Hien D, Kiba Koumare A, Barry N, Baguiya A, Hema A, Dianda F, Savadogo Y, Kouanda S, Tiono AB, Sirima SB. Protocol for a quasi-experimental study to assess the feasibility, acceptability and costs of multiple first-lines artemisinin-based combination therapies for uncomplicated malaria in the Kaya health district, Burkina Faso. BMJ Open. 2021 Feb 15;11(2):e040220. doi: 10.1136/bmjopen-2020-040220. PMID 33589447